CLINICAL TRIAL: NCT00228488
Title: Phase II Study of Iressa With/Without Concurrent Chemoradiotherapy in Patients With Advanced Non-Nasopharyngeal Head and Neck Carcinoma and to Study the Effect of Iressa™ (ZD1839) on Tumour Gene Expression Profiles ®
Brief Title: Effect of Iressa With/Without Concurrent Chemoradiotherapy on Tumor Gene Expression Profiles in Patients With Advanced Non-Nasopharyngeal Head and Neck Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1839IL/0547
Record Dates: First submitted 2005-09-27; First posted 2005-09-29 (Estimated); Last update posted 2007-12-19 (Estimated); Status verified 2007-12

CONDITIONS: Head and Neck Cancer
Keywords: advanced non-nasopharyngeal head and neck carcinoma
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Gefitinib

INTERVENTIONS:
Drug: Gefitinib

SUMMARY:
Two different patient populations will be targeted for this study. The first population (SP1) will include patients with recurrent/metastatic head and neck cancers, excluding salivary gland carcinomas. The second population (SP2) will include treatment-naïve patients with locally advanced squamous cell head and neck cancer (SCHNC).

SP1 will be treated with palliative intent and the patients can be treatment-naïve or have received prior chemotherapy. Study treatment will consist of Iressa (gefitinib) alone.

SP2 will be treated with radical intent. The patients must be treatment-naïve and study treatment will consist of induction Iressa for 3 weeks followed by a combination of Iressa plus cisplatin and concurrent irradiation.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed carcinoma of the head and neck (excluding salivary gland and nasopharyngeal carcinoma), namely squamous cell or undifferentiated carcinoma
* Recurrent/metastatic disease that is not amenable to cure
* Accessible tumour site for repeat tumour samplings
* Patients must be agreeable to repeated tumour samplings.
* Measurable disease sites by computed tomography (CT) imaging is preferred but not mandatory.
* Adequate performance status of ECOG 0 - 2
* Life expectancy of at least 3 months
* Written informed consent to participate in the study

Exclusion Criteria:

* Prior treatment with tyrosine kinase inhibitor or anti-epidermal growth factor receptor (EGFR) therapy
* Refusal for repeated tumour samplings
* Tumour site deemed unsafe for repeated samplings due to risk of bleeding
* In the opinion of the investigator, any evidence of severe or uncontrolled systemic disease (eg. unstable or uncompensated respiratory disorder, cardiac failure, hepatic decompensation, renal failure, uncontrolled metabolic disorders such as diabetes mellitus, or uncontrolled significant infections)
* Any bleeding disorders
* Pregnancy or breast-feeding (women of child-bearing potential)
* Other co-existing malignancies or malignancies diagnosed within the last 5 years with the exception of basal cell carcinoma or cervical carcinoma-in-situ

Inclusion Criteria for SP2:

* Histologically confirmed carcinoma of the head and neck (excluding salivary gland and nasopharyngeal carcinoma), namely squamous cell carcinoma or undifferentiated carcinoma
* Locally advanced disease (stage III/IV) without distant metastases, not amenable to curative resection, or patient refusal for surgery
* Accessible primary site for repeat tumour samplings
* Patients agreeable to repeated tumour samplings
* Evaluable and/or measurable disease sites on CT scans
* Adequate performance status of ECOG 0 - 1
* Written informed consent to participate in the study

Exclusion Criteria for SP2:

* Presence of distant metastases
* Prior treatment with EGFR-targeted therapy, or chemotherapy or radiotherapy to head and neck region
* Refusal for repeated tumour samplings
* Tumour site deemed unsafe for repeated samplings due to risk of bleeding
* Common toxicity criteria (CTC) grade 2 or greater pre-existing motor or sensory neuropathy
* In the opinion of the investigator, any evidence of severe or uncontrolled systemic disease (eg. unstable or uncompensated respiratory disorder, cardiac failure, hepatic decompensation, renal failure, uncontrolled metabolic disorders such as diabetes mellitus, or uncontrolled significant infections)
* Any bleeding disorders
* Absolute neutrophil count of less than 1000/mm3, and platelet count of less than 100,000/mm3
* Serum bilirubin greater than 2 times the upper limit of normal range (ULNR)
* Serum alanine aminotransferase (ALT) and serum aspartate amino transferase (AST) greater than 2.5 times ULNR
* Serum creatinine greater than 143 umol/litre
* Pregnancy or breast-feeding (women of child-bearing potential)
* Other co-existing malignancies or malignancies diagnosed within the last 5 years with the exception of basal cell carcinoma or cervical carcinoma-in-situ

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2004-06; Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
To study the effect of Iressa on gene expression profiles in patients with head and neck cancer

SECONDARY OUTCOMES:
To study the efficacy of Iressa as monotherapy as first line or after failing prior platinum-based regimen in patients with recurrent/metastatic head and neck carcinomas

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Medical Department, Study Director — AstraZeneca
Locations (2):
- Hong Kong, Hong Kong
- Singapore, Singapore